CLINICAL TRIAL: NCT03213405
Title: A Double Blind, Controlled by Conventional BCG, Dose-escalation Phase I Study, to Evaluate Safety, Tolerability and Immunogenicity of a Mycobacterium Bovis BCG (Bacillus Calmette-Guérin) Vaccine, 1331 Danish Strain, Live Attenuated and Recombinant for the Expression of Human Respiratory Syncytial Virus Nucleoprotein (N) in Healthy Males Within 18 and 50 Years of Age
Brief Title: A Study to Assess Safety, Tolerability and Immunogenicity of the Live Attenuated hRSV Vaccine rBCG-N-hRSV
Acronym: EVA-VRS01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government); Millennium Institute on Immunology and Immunotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-216; rBCG-N-VRSh 001 (Other: Instituto de Salud Pública de Chile)
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: human Respiratory Syncytial Virus; Phase I; Recombinant BCG vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional BCG full dose (Active Comparator): Participants will receive one full dose of the Conventional BCG vaccine administered as an intradermal injection at study entry.
  Interventions: Biological: Conventional BCG full dose
- rBCG-N-hRSV 1/100 dose (Experimental): Participants will receive one 1/100 dose of the rBCG-N-hRSV vaccine administered as an intradermal injection at study entry.
  Interventions: Biological: rBCG-N-hRSV 1/100
- rBCG-N-hRSV 1/10 dose (Experimental): Participants will receive one 1/10 dose of the rBCG-N-hRSV vaccine administered as an intradermal injection at study entry.
  Interventions: Biological: rBCG-N-hRSV 1/10
- rBCG-N-hRSV full dose (Experimental): Participants will receive one full dose of the rBCG-N-hRSV vaccine administered as an intradermal injection at study entry.
  Interventions: Biological: rBCG-N-hRSV full dose

INTERVENTIONS:
Biological: rBCG-N-hRSV 1/100 — 5x10^3 colony forming units (CFU) of rBCG-N-hRSV will be administered as an intradermal injection.
  Arms: rBCG-N-hRSV 1/100 dose
Biological: rBCG-N-hRSV 1/10 — 5x10^4 colony forming units (CFU) of rBCG-N-hRSV will be administered as an intradermal injection.
  Arms: rBCG-N-hRSV 1/10 dose
Biological: rBCG-N-hRSV full dose — 1x10^5 colony forming units (CFU) of rBCG-N-hRSV will be administered as an intradermal injection.
  Arms: rBCG-N-hRSV full dose
Biological: Conventional BCG full dose — 2x10^5 colony forming units (CFU) of conventional BCG will be administered as an intradermal injection.
  Arms: Conventional BCG full dose

SUMMARY:
Human respiratory syncytial virus (hRSV) is the main cause of lower respiratory tract infection in children under one year of age. This study will evaluate the safety, tolerability and immunogenicity of a recombinant Mycobacterium bovis BCG vaccine that expresses the human Respiratory Syncytial Virus Nucleoprotein (N), in adult males (18 to 50 years of age).

DETAILED DESCRIPTION:
hRSV is the main cause of infections in the lower respiratory tract, causing pneumonia, bronchiolitis and alveolitis in children younger than two years old. The infection is associated with the development of recurrent obstructive episodes in children with genetic predisposition. These hRSV infections also cause a high number of hospitalizations during the winter season.

At Pontificia Universidad Católica de Chile, a vaccine has been developed to prevent hRSV infection, which is the conventional Bacillus Calmette Guerin (BCG) vaccine modified to recombinantly express the Nucleoprotein of hRSV (rBCG-N-hRSV). This vaccine has proven to be safe and immunogenic in different animal models, both in Chile and the USA. Doses of this vaccine have been manufactured under Current Good Manufacturing Practices (cGMP) conditions in USA, which are suitable to be tested in humans. Due to the unique immunogenic and safety characteristics observed in animal models used to test the efficacy of the rBCG-N-hRSV vaccine prototype, this clinical study will evaluate safety, tolerability and immunogenicity of the immunogenic cGMP formulation in healthy adults.

Main objective: To characterize the safety and tolerability of escalating doses of the rBCG-N-hRSV vaccine, including doses of 5x10^3, 5x10^4 and 1x10^5 CFU (1%, 10% and 100% of the total dose) in healthy adult males of 18 to 50 years of age.

Secondary objectives:

1. To characterize the immune response against the Nucleoprotein of the hRSV in the previously stated escalating doses in the rBCG-N-hRSV.
2. To characterize the immune response against the Mycobacterium in the previously stated escalating doses in the rBCG-N-hRSV.

Study design: It corresponds to a phase I study, double blind (participant and personnel of the study) for the immunization of the tested vaccine or the control vaccine (Conventional BCG) within each cohort, to be performed in healthy adult males of 18 to 50 years of age.

After a full clinical and laboratory evaluation to discard diseases, immunodeficiencies and latent tuberculosis infection, the participants will be enrolled into three cohorts in a open and successive manner. Within each cohort, they will be randomly and in a blind-manner assigned to receive the tested vaccine (rBCG-N-hRSV) or the control vaccine (conventional BCG).

Cohort A: 6 participants vaccinated with 5x10^3 CFU of the rBCG-N-hRSV (1/100 part of the full dose) and 2 participants vaccinated with the conventional BCG (full dose).

Cohort B: 6 participants vaccinated with 5x10^4 CFU of the rBCG-N-hRSV (1/10 part of the full dose) and 2 participants vaccinated with the conventional BCG (full dose).

Cohort C: 6 participants vaccinated with 1x10^5 CFU of the rBCG-N-hRSV (full dose) and 2 participants vaccinated with the conventional BCG (full dose).

Each cohort will be completed within two weeks, followed by a period of 4 weeks of follow-up, in which the security data will be evaluated by a Data and Safety Monitoring Board (DSMB), who will determinate whether, according to the previously defined parameters, the escalation to the next cohort is possible, the cohort must be repeated, or whether the study must be stopped.

The DSMB is constituted by 5 physician experts in microbiology, virology/vaccinology and tuberculosis, with a wide national recognition, affiliated to institutions different from the sponsoring institution.

Number of participants: A minimum of 24 subjects, 8 by cohort. 18 participants will receive the tested vaccine and 6 will receive the control vaccine.

Main variables: Safety and tolerability.

* Evaluation of reactogenicity (Local and systemic Adverse Events-AE)
* Evaluation of laboratory AE
* Serious AE
* Evaluation of the presence of the vaccine in body fluids

Secondary variables: Immunogenicity

* Evaluation of the immune response against M. bovis BCG.
* Evaluation of the immune response against hRSV-N.

ELIGIBILITY:
Inclusion Criteria:

* Chilean male within 18 and 50 years old.
* To have accepted his voluntary participation through the sign of the informed consent.
* To be in good health, according to the medical history, physical examination and normal laboratory tests.
* To be vaccinated with BCG once or twice during his life.

Exclusion Criteria:

* Symptoms or diagnosis suggesting some systemic disease including renal, liver, cardiovascular or pulmonary impairment, immunodeficiency, autoimmune disease, malignancies, psychiatric or other conditions that can interfere on the interpretation of the results or compromise the health of the participants.
* Body mass index lower than 19 and higher that 30 kg/m2 and/or weight under 50 kg.
* Not being able to attend all the study visits (face-to-face and call phones) or not follow the specified instructions (fasting, not doing intense physical exercise during the previous 24 hours to the visits and 72 hours post-vaccine).
* Signs of latent or active infectious diseases by Mycobacterium tuberculosis (TB): QuantiFERON-TB positive test or Chest X-ray suggesting Tuberculosis (TBC).
* Positive screening for Human Immunodeficiency Virus (HIV), Hepatitis B superficial antigen (HBsAG) and anti-Hepatitis C Virus (HCV).
* Evidence of primary or secondary immunodeficiency, determined by history, physical test and levels of serum immunoglobulins and lymphocytes sub-populations at the screening.
* Use of immunosuppressors during the last 6 months previous to the visit.
* Use of inhaled corticosteroids during the last year or with antecedents of bronchial hyper-reactivity.
* Antecedents of intradomiciliary contact with subjects with Tuberculosis or other mycobacteria, even when he/she is under treatment.
* Antecedents of substance abuse (drugs or alcohol), according to DSM IV (See footnote*)
* Occurrence of any serious adverse event associated to the previous BCG vaccination.
* History of severe allergic reaction or anaphylaxis to vaccines
* History of severe infections (use of IV antibiotics, opportunist, latent TBC, herpes zoster) during six months previous to the visit.
* Not use or rejection to the use of contraceptives during the whole study (See footnote**).
* Administration of Immunoglobulins or blood-derived products during the six months previous to the visit or the planning of its use during the study.
* Eczema at the vaccination site (deltoid zone).
* Antecedents of keloid scar.
* Being vaccinated with BCG during the last 10 years.
* History of being vaccinated with BCG three or more times or the presence of three BCG scars.
* Using other investigational products during the 30 days previous to the study.
* Administration of any vaccine during the 8 weeks previous to the recruitment.
* Planned administration of any other different vaccine 30 days after the vaccination with the rBCG-N-hRSV.
* Acute illness symptoms and/or feverish symptoms at the time or during the last seven days previous to the recruitment (fever defined as an oral or axillary temperature of >38ºC).

(*) Substance abuse (drugs or alcohol): Maladaptive pattern of substance abuse that leads to a deterioration or clinical significant discomfort, expressed by one or more associated problems, during a time of twelve months, in one of the four vitals areas: inability to achieve main obligations; consume in dangerous situations, such as driving a vehicle; legal problems; consume despite the social and interpersonal difficulties associated.

(**) Given the remote possibility of negative effects produced by the vaccination in the sperm, the recruitment will be performed only to volunteers that are not planning of conceiving a child during the study duration. In each visit, the abstinence fulfillment will be checked or the use of effective contraceptive.

Eligibility criteria:

The eligibility of the volunteers will be performed if they fulfill the inclusion criteria and fulfill none of the mentioned exclusion criteria, also presenting all the normal screening study.

All the volunteers must sign the Informed consent approved by the Ethic Committee of the "Facultad de Medicina" of the "Pontificia Universidad Católica de Chile", before starting the first screening visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Kalergis, PhD, Study Director — Pontificia Universidad Catolica de Chile; Katia Abarca, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bueno SM, Gonzalez PA, Cautivo KM, Mora JE, Leiva ED, Tobar HE, Fennelly GJ, Eugenin EA, Jacobs WR Jr, Riedel CA, Kalergis AM. Protective T cell immunity against respiratory syncytial virus is efficiently induced by recombinant BCG. Proc Natl Acad Sci U S A. 2008 Dec 30;105(52):20822-7. doi: 10.1073/pnas.0806244105. Epub 2008 Dec 15. PMID 19075247
- [Background] Cautivo KM, Bueno SM, Cortes CM, Wozniak A, Riedel CA, Kalergis AM. Efficient lung recruitment of respiratory syncytial virus-specific Th1 cells induced by recombinant bacillus Calmette-Guerin promotes virus clearance and protects from infection. J Immunol. 2010 Dec 15;185(12):7633-45. doi: 10.4049/jimmunol.0903452. Epub 2010 Nov 17. PMID 21084664
- [Background] Cespedes PF, Bueno SM, Ramirez BA, Gomez RS, Riquelme SA, Palavecino CE, Mackern-Oberti JP, Mora JE, Depoil D, Sacristan C, Cammer M, Creneguy A, Nguyen TH, Riedel CA, Dustin ML, Kalergis AM. Surface expression of the hRSV nucleoprotein impairs immunological synapse formation with T cells. Proc Natl Acad Sci U S A. 2014 Aug 5;111(31):E3214-23. doi: 10.1073/pnas.1400760111. Epub 2014 Jul 23. PMID 25056968
- [Background] Palavecino CE, Cespedes PF, Gomez RS, Kalergis AM, Bueno SM. Immunization with a recombinant bacillus Calmette-Guerin strain confers protective Th1 immunity against the human metapneumovirus. J Immunol. 2014 Jan 1;192(1):214-23. doi: 10.4049/jimmunol.1300118. Epub 2013 Dec 6. PMID 24319265
- [Background] Cespedes PF, Rey-Jurado E, Espinoza JA, Rivera CA, Canedo-Marroquin G, Bueno SM, Kalergis AM. A single, low dose of a cGMP recombinant BCG vaccine elicits protective T cell immunity against the human respiratory syncytial virus infection and prevents lung pathology in mice. Vaccine. 2017 Feb 1;35(5):757-766. doi: 10.1016/j.vaccine.2016.12.048. Epub 2017 Jan 5. PMID 28065474
- [Derived] Pacheco GA, Andrade CA, Galvez NMS, Vazquez Y, Rodriguez-Guilarte L, Abarca K, Gonzalez PA, Bueno SM, Kalergis AM. Characterization of the humoral and cellular immunity induced by a recombinant BCG vaccine for the respiratory syncytial virus in healthy adults. Front Immunol. 2023 Jul 18;14:1215893. doi: 10.3389/fimmu.2023.1215893. eCollection 2023. PMID 37533867
- [Derived] Abarca K, Rey-Jurado E, Munoz-Durango N, Vazquez Y, Soto JA, Galvez NMS, Valdes-Ferrada J, Iturriaga C, Urzua M, Borzutzky A, Cerda J, Villarroel L, Madrid V, Gonzalez PA, Gonzalez-Aramundiz JV, Bueno SM, Kalergis AM. Safety and immunogenicity evaluation of recombinant BCG vaccine against respiratory syncytial virus in a randomized, double-blind, placebo-controlled phase I clinical trial. EClinicalMedicine. 2020 Oct 6;27:100517. doi: 10.1016/j.eclinm.2020.100517. eCollection 2020 Oct. PMID 33073219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed in a single center. Recruitment started on 06.27.17 and ended on 12.04.17.
Period: Overall Study
Arm/Group | Conventional BCG Full Dose | rBCG-N-hRSV 1/100 Dose | rBCG-N-hRSV 1/10 Dose | rBCG-N-hRSV Full Dose
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional BCG Full Dose | rBCG-N-hRSV 1/100 Dose | rBCG-N-hRSV 1/10 Dose | rBCG-N-hRSV Full Dose | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 22.0 [19 to 31] | 28.5 [21 to 36] | 24.0 [22 to 44] | 21.0 [20 to 25] | 23.875 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Chile | 6 | 6 | 6 | 6 | 24
Previously vaccinated with BCG [Count of Participants; unit: Participants] | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Required Adverse Events Grade II, III, and IV, Laboratory Adverse Events Grade II, III, and IV, and Severe Considered Adverse Events Related to the Vaccine.
Description: To determine the safety of the rBCG-N-hRSV by evaluating the number of vaccinated participants with adverse events (AEs) due to the vaccination. Among these AEs, the following will be measured: Number of subjects with required AEs grade II, III, and IV, laboratory AEs grade II, III, and IV, and severe AEs (SAEs) considered related to the vaccine.
  Required AEs included pain, induration, pustule, fever, headache, myalgia, and diarrhea, among others. AEs were collected by self-report on diary cards, study visits, and study phone calls.
  Laboratory AEs included hematological and biochemical parameters, such as blood counts, transaminases, cholesterol, creatine phosphokinase, and urine analyses, among others.
  SAEs were defined as any untoward medical occurrence that resulted in death; was life-threatening; required hospitalization; or resulted in disability, among others. Grade 4 laboratory AEs were also considered SAEs.
Time Frame: Up to 180 days post-vaccination (A total of 11 months and 6 days for the whole study)
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional BCG Full Dose | rBCG-N-hRSV 1/100 Dose | rBCG-N-hRSV 1/10 Dose | rBCG-N-hRSV Full Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Required adverse events grade II | 6 | 6 | 6 | 6
  Required adverse events grade III | 0 | 0 | 0 | 1
  Required adverse events grade IV | 0 | 0 | 0 | 0
  Laboratory adverse events grade II | 3 | 5 | 2 | 4
  Laboratory adverse events grade III | 2 | 1 | 2 | 1
  Laboratory adverse events grade IV | 1 | 0 | 0 | 0
  Severe adverse events related to the vaccine | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 180 days post-vaccination (A total of 11 months and 6 days for the whole study).
Description: Participants received a single dose of the vaccine, administered intradermally in the deltoid area following the standard national protocol for BCG vaccination used in Chile, and were observed during the following 3 hours. Participants were then evaluated at 1-3, 7, 14, 30, 60, 120, and 180 days post-vaccination. Follow up phone calls were performed at 4, 21, 45, 90, and 150 dpv.
Arm/Group | Conventional BCG Full Dose | rBCG-N-hRSV 1/100 Dose | rBCG-N-hRSV 1/10 Dose | rBCG-N-hRSV Full Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional BCG Full Dose (N=6) | rBCG-N-hRSV 1/100 Dose (N=6) | rBCG-N-hRSV 1/10 Dose (N=6) | rBCG-N-hRSV Full Dose (N=6)
Increase in CPK (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — A grade 4 increase in CPK 15 days after vaccination with the control BCG, related to intense physical exercise two days before the exam. CPK values returned to normal levels in an analysis performed 16 days later
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional BCG Full Dose (N=6) | rBCG-N-hRSV 1/100 Dose (N=6) | rBCG-N-hRSV 1/10 Dose (N=6) | rBCG-N-hRSV Full Dose (N=6)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased CPK (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocyturia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased aspartate aminotransferase (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pustule at the inoculation site (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Scab at the inoculation site (General disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Sensitivity at the inoculation site (General disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2)
Erythema at the inoculation site (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Induration at the inoculation site (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 6 (13) | 6 (8) | 2 (2) | 6 (7)
Fatigue (General disorders) | 2 (2) | 3 (6) | 2 (3) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (7) | 2 (3) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (6) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Hypertension (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hypotension (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03213405/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT03213405/ICF_001.pdf